CLINICAL TRIAL: NCT03510455
Title: BGJ398 for the Treatment of Tumor-Induced Osteomalacia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was stopped early due to a greater than expected incidence of ocular AEs and analysis of the data from the first 4 subjects indicating that the likelihood of permanent remission with this therapy was low.
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180086; 18-D-0086
Record Dates: First submitted 2018-04-26; First posted 2018-04-27 (Actual); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2020-05

CONDITIONS: Tumor-Induced Osteomalacia; Oncogenic Osteomalacia
Keywords: FGF-23; Fibroblast Growth Factor (FGF23); Hypophosphatemia
MeSH Terms: conditions — Oncogenic osteomalacia; Hypophosphatemia | interventions — infigratinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (TIO Subjects) (Experimental): Phase 2, open-label, non-randomized, single-arm, drug treatment trial. 10 subjects will be studied. Treatment duration of 6 months with 3 months off drug follow-up and optional extension phase.
  Interventions: Drug: BGJ398

INTERVENTIONS:
Drug: BGJ398 — BGJ398, a pan-fibroblast growth factor receptor (FGFR) kinase inhibitor will be orally administered over six 4-week cycles (4 weeks on drug continuously). After the initial dose, escalation/de- escalation of BGJ398 will be based on FGF- 23 blood levels and adjusted according to protocol procedures. The six cycles of BGJ398 will be followed by 3 months off the drug and an optional extension phase.

SUMMARY:
Background:

People with tumor-induced osteomalacia (TIO) have small tumors that may cause low blood phosphorus, weak muscles, bone pain, and broken bones. The tumors may be so small they are hard to find or impossible to remove. Researchers want to test a drug that may help treat TIO.

Objective:

To see how the drug BGJ398 affects people with tumor-induced osteomalacia.

Eligibility:

People ages 18-85 who are in NIH protocol 01-D-0184 and have TIO that cannot be found or easily removed

Design:

At every study visit, participants will have:

* Medical history
* Physical exam
* Blood and urine tests
* Questions about their health and fatigue

At the screening visit, participants will also have a heart and eye tests. They may have other tests to find their tumor.

The baseline visit will be a 1-week stay in the clinic. Participants will have the regular study tests, plus:

* Their first dose of the study drug capsules
* Blood and urine collected every 2-4 hours for 24 hours. A thin plastic tube will be inserted in a vein to collect blood.
* Heart and kidney ultrasounds
* Activities that test strength
* 6-minute walk test

Participants will take the study drug for six 1-month cycles. In each cycle, participants will:

* Take the study drug every day for 4 weeks.
* Have 1 visit. Participants will collect their urine for 24 hours and have their blood drawn. Participants will have the regular study tests and repeat some baseline tests.
* Have blood and urine tests at their local lab.

Participants will have 1 visit at the end of the last cycle and another 3 months later....

DETAILED DESCRIPTION:
Background:

* Tumor-induced osteomalacia (TIO) is a rare disorder in which fibroblast growth factor (FGF23)-producing neoplasms cause renal phosphate wasting and skeletal disease.
* Recent studies have shown that chromosomal translocations causing a fibronectin-FGFR1 (FN1/FGFR1) fusion gene have been identified in 40-60% of these tumors.
* BGJ398 is an orally bio-available, selective and ATP competitive pan-fibroblast growth factor receptor (FGFR) kinase inhibitor which has demonstrated anti-tumor activity in preclinical, in vitro and in-vivo tumor models harboring FGFR genetic alterations.

Objectives:

To induce complete metabolic response in subjects with tumor-induced osteomalacia (TIO) with BGJ-398 as demonstrated by normalization of FGF23 and phosphate homeostasis.

Eligibility:

Patients may be eligible if they:

* Are adults 18-85 years with documented evidence of TIO due to a non-localized or unresectable tumor, or metastatic disease, or resectable tumor that cannot be easily removed.
* Are not taking any exclusionary medications or foods that may interfere with BGJ398.
* Are not pregnant or nursing and are willing to use contraception (at least two forms of contraception), if able to become pregnant.
* Have no significant ophthalmologic, gastrointestinal, renal, or hematologic disease.

Design:

* Phase 2, open-label, non-randomized, single-arm, drug treatment trial.
* 10 subjects to be studied.
* Treatment duration 6 months with 3 months off drug follow-up and optional extension phase.
* Monthly NIH visits with additional labs obtained in between visits.
* Imaging performed in those with identifiable tumors.
* Analyses to include repeated measures ANOVA assessing changes in biochemical indices over time in response to BGJ398.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients eligible for inclusion in this study have to meet all of the following criteria:

* Aged 18-85 years
* Diagnosis of TIO due to a non-localized or unresectable tumor, or metastatic disease or resectable tumor that cannot be removed by minor surgical procedure. This diagnosis will be confirmed prior to enrollment on protocol 01-D-0184. Where clinically indicated, genetic testing to rule-out heritable causes of FGF23 excess will also be performed on 01-D-0184.
* Willing and able to comply with scheduled visits, treatment plan and laboratory tests.
* Able to swallow and retain oral medication.
* Able to provide informed consent

EXCLUSION CRITERIA:

Patients eligible for this study must not meet any of the following criteria:

* Have another genetic or secondary cause of hypophosphatemia.
* History of any other malignancy that has not been cured/in remission for 5 years.
* Patients who previously received treatment with an FGFR inhibitor other than BGJ398.
* Current evidence of corneal or retinal disorder/keratopathy including, but not limited to: bullous/band keratopathy, corneal abrasion, inflammation/ulceration, keratoconjuctivitis, confirmed by ophthalmologic examination
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral BGJ398 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection)
* Patients who are currently receiving treatment with agents that are known strong inducers or inhibitors of CYP3A4 are prohibited. This includes treatment with enzyme-inducing antiepileptic drugs including carbamazepine, phenytoin, phenobarbital, and primidone.
* Consumption of grapefruit, grapefruit juice, pomegranates, star fruits, Seville oranges or products within 7 days prior to first dose
* Use of amiodarone within 90 days prior to first dose
* Current use of therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulants. Heparin and/or low molecular weight heparins are allowed.
* Insufficient bone marrow function defined as all of the following:

  * ANC <1,500/mm^3 [1.0 x 10^9/L] AND
  * Platelets < 75,000/mm^3 [75 x 10^9/L] AND
  * Hemoglobin < 10.0 g/dL
* Insufficient hepatic and renal function defined as one of the following:

  * Total bilirubin > 1.5x ULN OR
  * AST/SGOT and ALT/SGPT > 2x ULN OR
  * Blood creatinine > 1.5xULN and/or calculated eGFR < 45 ml/min/1.73 m^2 (calculated by CKD-Epi)
* Clinically significant cardiac disease including any of the following:

  * Congestive heart failure requiring treatment (NY Heart Association grade >= 2),
  * History or presence of clinically significant ventricular arrhythmias, atrial fibrillation, resting bradycardia, or conduction abnormality
  * Unstable angina pectoris or acute myocardial infarction less than or equal to 3 months prior to starting study drug
  * QTcF > 450 msec (males); > 470 msec (females)
  * History of congenital long QT syndrome
* Recent (less than or equal to 3 months) transient ischemic attack or stroke
* Patients under age 21 will have a bone age assessed as part of their clinically indicated skeletal survey under 01-D-0184 and will not be offered enrollment if their growth plates are open.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 3 months following the discontinuation of study treatment. Highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male sterilization (at least 6 months prior to screening). For female subjects on the study the vasectomized male partner should be the sole partner for that subject.
  * Combination of the following (a+b or a+c, or b+c):

    * Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception
    * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository

      * Post-menopausal women are allowed to participate in this study. Women are considered post- menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH >40 mIU/ml or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
      * Sexually active males unless they use a condom during intercourse while taking drug and for 3 months after the last dose of the study drug and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
      * Patients with TIO who are currently taking BGJ398 or have been treated with BGJ398 in the past are eligible to participate in this study, provided that they discontinue BGJ398 for 2 weeks prior to the baseline visit.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel I Gafni, M.D., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-D-0086.html

RESULTS

PARTICIPANT FLOW:
Groups:
- TIO Subjects Who Received BGJ398 (Single Arm): TIO subjects were treated with BGJ398 for 24 weeks with optional extension phase
Period: Overall Study
Arm/Group | TIO Subjects Who Received BGJ398 (Single Arm)
Started | 4
Treated | 4
Extension Phase | 1
Screening Failures | 0
Completed | 3 (3 of 4 patients completed the 24 week treatment phase of the study)
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Single Arm (TIO Subjects): Phase 2, open-label, non-randomized, single-arm, drug treatment trial. 10 subjects will be studied. Treatment duration of 6 months with 3 months off drug follow-up and optional extension phase.
  BGJ398: BGJ398, a pan-fibroblast growth factor receptor (FGFR) kinase inhibitor will be orally administered over six 4-week cycles (3 weeks on drug, 1 week off drug). After the initial dose, escalation/de- escalation of BGJ398 will be based on FGF- 23 blood levels and adjusted according to protocol procedures. The six cycles of BGJ398 will be followed by 3 months off the drug and an optional extension phase.
Arm/Group | Single Arm (TIO Subjects)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.75 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Type of TIO Disease [Count of Participants; unit: Participants]
  Localized | 2
  Non-localized | 2
  Metastatic | 0
Blood Intact FGF23 on Initiation of Sutdy [Mean (Standard Deviation); unit: pg/mL] | 1384 (1467)
Blood C-Terminal FGF23 on Initiation of Study [Mean (Standard Deviation); unit: RU/mL] | 814 (911)
Blood Phosphate on Initiation of Study [Mean (Standard Deviation); unit: mg/dL] | 1.6 (0.3)
Blood Alkaline Phosphatase on Initiation of Study [Mean (Standard Deviation); unit: U/L] | 134 (54)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Metabolic Remission After Stopping BGJ398
Description: Participants were monitored for up to 12 weeks after stopping BGJ398. A participant was considered to have a complete metabolic remission by achieving both normal blood FGF23 and phosphorus levels in the blood for 12 weeks after stopping BGJ398.
Time Frame: Up to 12 weeks after stopping BGJ398
Population: The population consisted of all participants enrolled in the study
Measure: Count of Participants; unit: Participants
Arm/Group | TIO Subjects Who Received BGJ398 (Single Arm)
Number analyzed (Participants) | 4
Participants
  Complete Metabolic Remission | 0
  No Complete Metabolic Remission | 4

2. Secondary Outcome: Number of Participants With Complete and Partial Metabolic Response Rate
Description: Participants were monitored for metabolic response to BGJ398 every other week. A participant was considered to have a complete metabolic response by achieving both normal c-terminal FGF23 and phosphorus levels at each time point. A participant was considered to have a partial metabolic response by achieving both a decrease of at least 50% in c-terminal FGF23 levels and an increase of at least 50% in phosphorous at each time point
Time Frame: Every 2 weeks up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm (TIO Subjects)
Number analyzed (Participants) | 4
Participants
  Baseline: Complete Metabolic Response | 0
  Baseline: Partial Metabolic Response | 0
  Baseline: Neither Complete or Partial Metabolic Response | 4
  Week 2: Complete Metabolic Response | 2
  Week 2: Partial Metabolic Response | 1
  Week 2: Neither Complete or Partial Metabolic Response | 1
  Week 4: Complete Metabolic Response | 0
  Week 4: Partial Metabolic Response | 1
  Week 4: Neither Complete or Partial Metabolic Response | 3
  Week 6: Complete Metabolic Response | 2
  Week 6: Partial Metabolic Response | 1
  Week 6: Neither Complete or Partial Metabolic Response | 1
  Week 8: Complete Metabolic Response | 1
  Week 8: Partial Metabolic Response | 1
  Week 8: Neither Complete or Partial Metabolic Response | 2
  Week 10: Complete Metabolic Response | 0
  Week 10: Partial Metabolic Response | 0
  Week 10: Neither Complete or Partial Metabolic Response | 4
  Week 12: Complete Metabolic Response | 1
  Week 12: Partial Metabolic Response | 1
  Week 12: Neither Complete or Partial Metabolic Response | 2
  Week 14: Complete Metabolic Response | 1
  Week 14: Partial Metabolic Response | 1
  Week 14: Neither Complete or Partial Metabolic Response | 2
  Week 16: Complete Metabolic Response | 0
  Week 16: Partial Metabolic Response | 1
  Week 16: Neither Complete or Partial Metabolic Response | 3
  Week 18: Complete Metabolic Response | 1
  Week 18: Partial Metabolic Response | 2
  Week 18: Neither Complete or Partial Metabolic Response | 1
  Week 20: Complete Metabolic Response | 1
  Week 20: Partial Metabolic Response | 1
  Week 20: Neither Complete or Partial Metabolic Response | 2
  Week 22: Complete Metabolic Response | 1
  Week 22: Partial Metabolic Response | 1
  Week 22: Neither Complete or Partial Metabolic Response | 2
  Week 24 - prior to drug discontinuation: Complete Metabolic Response | 0
  Week 24 - prior to drug discontinuation: Partial Metabolic Response | 0
  Week 24 - prior to drug discontinuation: Neither Complete or Partial Metabolic Response | 4
  Week 24 - after drug discontinuation: Complete Metabolic Response | 0
  Week 24 - after drug discontinuation: Partial Metabolic Response | 0
  Week 24 - after drug discontinuation: Neither Complete or Partial Metabolic Response | 4

3. Secondary Outcome: Number of Participants With Grade 3 or 4 Adverse Events or Serious Adverse Events
Description: Percentage of patients who incurred grade 3 or 4 adverse events (AEs) or serious adverse events (SAE) or AEs causing dose interruption/reduction
Time Frame: 24 week treatment phase followed by 3 month follow up or extension phase
Measure: Count of Participants; unit: Participants
Arm/Group | TIO Subjects Who Received BGJ398 (Single Arm)
Number analyzed (Participants) | 4
Participants
  SAE | 0
  Grade 4 AE | 0
  Grade 3 AE | 1
  AE leading to dose interruption/reduction | 4

4. Secondary Outcome: Six-Minute Walk Test
Description: The Six-Minute Walk Test (6MWT), is a self-paced practical test that measures the distance the patient can quickly cover on a flat, hard surface. Each subject was instructed to complete the maximum distance possible in six minutes. Feedback was given in two minute intervals and during the last 30 seconds. Patients were instructed to notify test administrator of leg cramping, pain, nausea, dizziness and shortness of breath. Test administrators counted each lap and upon test completion, the partial distance is measured and added to where the subject stopped.
Time Frame: Assessed at baseline and 24 weeks after starting BGJ398
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | TIO Subjects Who Received BGJ398 (Single Arm)
Number analyzed (Participants) | 4
Meters
  Baseline | 320.4 (221.8)
  24 Weeks | 496 (173.4)

5. Secondary Outcome: Hand Grip Strength Test
Description: The person is seated, lower extremities flexed at 90 degrees. The individual uses the dominant hand for this activity. The individual sit with shoulder adducted and neutrally rotated elbow flexed at 90 degrees, forearm in neutral position, resting on the arm of a chair. The JAMAR Hand Dynamometer set to the third level position from the inside is used. The examiner lightly supports the readout dial to prevent it from dropping. The patient is asked to "Squeeze as hard as you can….squeeze…..squeeze….relax." Three successive trials is recorded in kilograms. A 10-15 second break occurs to prevent muscle fatigue. Scores are recorded and averaged for the final result. Scores within two standard deviations of the mean are considered within normal limits.
Time Frame: Assessed at baseline and every 4 weeks up to 24 weeks during the treatment phase, and every 4 weeks in the follow up phase, up to 37 weeks
Population: Only 2 patients performed strength testing at 28 weeks.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | TIO Subjects Who Received BGJ398 (Single Arm)
Number analyzed (Participants) | 4
kg
  Baseline | 14.7 (11.8)
  Week 4 | 16.4 (11.2)
  Week 8 | 18.5 (9.4)
  Week 12 | 17.0 (7.9)
  Week 16 | 22.6 (18.5)
  Week 20 | 17.3 (6.6)
  Week 24 | 15.5 (1.4)
  Week 28: number analyzed (Participants) | 2
  Week 28 | 30.1 (6.7)

6. Secondary Outcome: Pinch Test
Description: A lateral pinch is required of the patient, using the dominant hand. The individual is seated, lower extremities flexed at 90 degrees. The examiner stabilizes the patient's wrist as the patient holds the pinch gauge to perform the test. The examiner requests the person to pinch with maximum strength. The peak-hold needle will automatically record the highest force exerted. After the patient uses the Pinch gauge, the examiner records the reading and resets the peak-hold needle to zero before testing again. Three lateral pinch trials are recorded and averaged for the final result.
Time Frame: Assessed at baseline and every 4 weeks for the 24 treatment period, and every 4 weeks in the follow up phase, up to 37 weeks
Population: Only 2 patients performed strength testing at 28 weeks.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | TIO Subjects Who Received BGJ398 (Single Arm)
Number analyzed (Participants) | 4
kg
  Baseline | 6.8 (4.0)
  Week 4 | 6.7 (1.2)
  Week 8 | 6.8 (1.3)
  Week 12 | 7.5 (2.0)
  Week 16 | 7.5 (1.0)
  Week 20 | 7.7 (1.5)
  Week 24 | 7.0 (1.3)
  Week 28: number analyzed (Participants) | 2
  Week 28 | 8.1 (1.9)

7. Secondary Outcome: Five Times Sit-to-Stand Test
Description: The Five Times Sit to Stand Test measures an aspect of transfer skill. The test provides a method to quantify functional lower extremity strength and/or identify movement strategies a patient uses to complete transitional movements.
  The chair is free standing. Patient sits with arms folded across chest and with their back against the chair. A standard chair height 44 cm was used for each patient. Patient stands fully between repetitions of the test, careful to not touch the back of the chair during each repetition. Patient instructions: "I want you to stand up and sit down 5 times as quickly as you can when I say Go." Timing begins at "Go" and ends when the buttocks touches the chair after the 5th repetition. The results are recorded in seconds.
Time Frame: Assessed at baseline and every 4 weeks during the 24 week treatment period
Population: Only 2 patients performed strength testing at 28 weeks.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | TIO Subjects Who Received BGJ398 (Single Arm)
Number analyzed (Participants) | 4
seconds
  Baseline | 14.7 (6.5)
  Week 4 | 13.2 (4.0)
  Week 8 | 13.5 (1.1)
  Week 12 | 11.2 (0.7)
  Week 16 | 10.5 (1.5)
  Week 20 | 10.8 (0.8)
  Week 24 | 11.1 (0.8)
  Week 28: number analyzed (Participants) | 2
  Week 28 | 11.1 (1.0)

8. Secondary Outcome: The Disabilities of Arm Shoulder and Hand Outcome Measurement (DASH)
Description: The Disabilities of Arm Shoulder and Hand Outcome Measurement (DASH) The minimum score value is 0, maximum is 100, where a higher school represents a worse outcome (significant symptoms/disability)
Time Frame: as for outcome 5
Population: 2 patients did not fill out their DASH at week 28
Measure: Mean (Standard Deviation); unit: DASH Disability/Symptom Score
Arm/Group | TIO Subjects Who Received BGJ398 (Single Arm)
Number analyzed (Participants) | 4
DASH Disability/Symptom Score
  Baseline | 16.5 (4.8)
  Week 4 | 13.3 (6.8)
  Week 8 | 14.2 (4.6)
  Week 12 | 13.3 (7.3)
  Week 16 | 12.7 (6.7)
  Week 20 | 21.0 (23.1)
  Week 24 | 12.1 (8.1)
  Week 28: number analyzed (Participants) | 2
  Week 28 | 10.0 (2.3)

9. Secondary Outcome: RAND SF-36 Survey Results
Description: Evaluation using the RAND 36-Item Short Form Survey (SF-36). Results were separated into 8 domains - Physical Functioning, Role limitations due to physical health problems, Role limitations due to emotional problems, Emotional well-being, Energy/fatigue, Social functioning, Bodily Pain, and General health perceptions.
  The minimum value is 0, the maximum value is 100, which the higher the score, the better the outcome.
Time Frame: as for outcome 5
Population: Only 2 patients completed week 28 surveys
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TIO Subjects Who Received BGJ398 (Single Arm)
Number analyzed (Participants) | 4
score on a scale
  Physical Functioning - Baseline | 46.3 (18.9)
  Physical Functioning - 4 weeks | 47.5 (21.0)
  Physical Functioning - 8 weeks | 51.3 (16.5)
  Physical Functioning - 12 weeks | 47.5 (12.6)
  Physical Functioning - 16 weeks | 56.0 (16.2)
  Physical Functioning - 20 weeks | 52.5 (26.0)
  Physical Functioning - 24 weeks | 41.0 (6.4)
  Physical Functioning - 28 weeks: number analyzed (Participants) | 2
  Physical Functioning - 28 weeks | 65.0 (7.1)
  Role limitations due to physical health problems - Baseline | 43.8 (12.5)
  Role limitations due to physical health problems - 4 weeks | 93.8 (12.5)
  Role limitations due to physical health problems - 8 weeks | 68.8 (31.5)
  Role limitations due to physical health problems - 12 weeks | 50 (35.4)
  Role limitations due to physical health problems - 16 weeks | 50 (57.7)
  Role limitations due to physical health problems - 20 weeks | 75 (50)
  Role limitations due to physical health problems - 24 weeks | 25 (50)
  Role limitations due to physical health problems - 28 weeks: number analyzed (Participants) | 2
  Role limitations due to physical health problems - 28 weeks | 12.5 (17.7)
  Role limitations due to emotional problems - Baseline | 66.7 (27.2)
  Role limitations due to emotional problems - 4 weeks | 83.3 (33.3)
  Role limitations due to emotional problems - 8 weeks | 75 (31.9)
  Role limitations due to emotional problems - 12 weeks | 66.7 (47.1)
  Role limitations due to emotional problems - 16 weeks | 50 (43)
  Role limitations due to emotional problems - 20 weeks | 91.7 (16.7)
  Role limitations due to emotional problems - 24 weeks | 41.7 (50)
  Role limitations due to emotional problems - 28 weeks: number analyzed (Participants) | 2
  Role limitations due to emotional problems - 28 weeks | 33.3 (47.1)
  Emotional well-being - Baseline | 67 (15.1)
  Emotional well-being - 4 weeks | 72 (15.7)
  Emotional well-being - 8 weeks | 72 (12.6)
  Emotional well-being - 12 weeks | 72 (17.6)
  Emotional well-being - 16 weeks | 69.8 (21.5)
  Emotional well-being - 20 weeks | 73 (8.2)
  Emotional well-being - 24 weeks | 62 (10.1)
  Emotional well-being - 28 weeks: number analyzed (Participants) | 2
  Emotional well-being - 28 weeks | 72 (5.7)
  Energy/fatigue - Baseline | 50 (29.4)
  Energy/fatigue - Week 4 | 58.8 (8.5)
  Energy/fatigue - week 8 | 52.5 (22.2)
  Energy/fatigue - week 12 | 46.3 (28.4)
  Energy/fatigue - week 16 | 61.3 (31.5)
  Energy/fatigue - week 20 | 57.5 (18.5)
  Energy/fatigue - week 24 | 48.8 (33.3)
  Energy/fatigue - week 28: number analyzed (Participants) | 2
  Energy/fatigue - week 28 | 47.5 (53.0)
  Social functioning - Baseline | 59.4 (37.3)
  Social functioning - 4 weeks | 87.5 (14.4)
  Social functioning - 8 weeks | 78.1 (21.3)
  Social functioning - 12 weeks | 81.3 (16.1)
  Social functioning - 16 weeks | 75 (27)
  Social functioning - 20 weeks | 78.1 (25.8)
  Social functioning - 24 weeks | 71.9 (32.9)
  Social functioning - 28 weeks: number analyzed (Participants) | 2
  Social functioning - 28 weeks | 75 (17.7)
  Bodily Pain - Baseline | 51.9 (29.2)
  Bodily Pain - week 4 | 66.3 (28)
  Bodily Pain - week 8 | 63.1 (37.4)
  Bodily Pain - week 12 | 43.1 (26.8)
  Bodily Pain - week 16 | 72.5 (34.6)
  Bodily Pain - week 20 | 75 (20.7)
  Bodily Pain - week 24 | 36.2 (2.5)
  Bodily Pain - week 28: number analyzed (Participants) | 2
  Bodily Pain - week 28 | 90 (0)
  General health perceptions - Baseline | 60 (10.8)
  General health perceptions - week 4 | 68.8 (13.1)
  General health perceptions - week 8 | 72.5 (16.6)
  General health perceptions - week 12 | 73.8 (25.9)
  General health perceptions - week 16 | 71.3 (14.9)
  General health perceptions - week 20 | 67.5 (23.3)
  General health perceptions - week 24 | 71.3 (18.0)
  General health perceptions - week 28: number analyzed (Participants) | 2
  General health perceptions - week 28 | 67.5 (31.8)

10. Secondary Outcome: PROMIS Fatigue
Description: Assessed using the PROMIS (Patient-Reported Outcomes Measurement Information System) Fatigue 8A short form.
  Scores are given as T values when compared to a population where the mean is 50 and 1SD is 10.
  A higher score represents increased feelings of fatigue.
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | TIO Subjects Who Received BGJ398 (Single Arm)
Number analyzed (Participants) | 4
T score
  Baseline | 55.1 (8.1)
  Week 4 | 47.4 (1.6)
  Week 8 | 52.6 (7.9)
  Week 12 | 52.3 (9.1)
  Week 16 | 52.3 (9.1)
  Week 20 | 46.6 (9.1)
  Week 24 | 52 (4.9)
  Week 28 | 46.7 (8.1)

11. Secondary Outcome: PROMIS Pain Interference Score
Description: Assessed using the PROMIS (Patient-Reported Outcomes Measurement Information System) Pain Interference 8A short form.
  Scores are given as T values when compared to a population where the mean is 50 and 1SD is 10.
  A higher score represents increased pain interference
Time Frame: as for outcome 5
Population: Only 2 patients completed the week 28 surveys
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | TIO Subjects Who Received BGJ398 (Single Arm)
Number analyzed (Participants) | 4
T score
  Baseline | 56.4 (4.5)
  Week 4 | 52.6 (9.4)
  Week 8 | 52.5 (6.0)
  Week 12 | 55.7 (4.2)
  Week 16 | 49.0 (10.6)
  Week 20 | 48.2 (15)
  Week 24 | 52.6 (9.1)
  Week 28: number analyzed (Participants) | 2
  Week 28 | 40.7 (0)

12. Secondary Outcome: PROMIS Mobility Score
Description: Assessed using the PROMIS (Patient-Reported Outcomes Measurement Information System) Mobility bank.
  Scores are given as T values when compared to a population where the mean is 50 and 1SD is 10.
  A higher score represents a better outcome (unencumbered mobility)
Time Frame: as for outcome 5
Population: Only 2 patients completed the week 28 surveys
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | TIO Subjects Who Received BGJ398 (Single Arm)
Number analyzed (Participants) | 4
T score
  Baseline | 38.2 (6.7)
  Week 4 | 40.0 (6.4)
  Week 8 | 39.3 (5.3)
  Week 12 | 38.8 (3.2)
  Week 16 | 40.2 (4.5)
  Week 20 | 40.7 (7.3)
  Week 24 | 39.5 (2.6)
  Week 28: number analyzed (Participants) | 2
  Week 28 | 43.6 (1.6)

13. Secondary Outcome: Blood Intact FGF23 Levels
Description: Measured Blood Intact FGF23 Levels.
Time Frame: Assessed at baseline and every 2 weeks up to 24 weeks during the treatment phase, and every 4 weeks in the follow up phase, up to 37 weeks
Population: There were dose interruptions throughout the 24 week treatment phase for 3 of the 4 subjects. Only 3 patients provided follow up samples.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | TIO Subjects Who Received BGJ398 (Single Arm)
Number analyzed (Participants) | 4
pg/mL
  Baseline | 1384 (1467)
  4 Weeks | 282 (254)
  8 Weeks | 286 (236)
  12 Weeks | 596 (924)
  16 Weeks | 310 (202)
  20 Weeks | 135 (67)
  24 Weeks | 439 (230)
  Follow up: number analyzed (Participants) | 3
  Follow up | 2534.8 (2824.6)

14. Secondary Outcome: Blood C-terminal FGF23 Level
Time Frame: as for outcome 13
Population: There were dose interruptions throughout the 24 week treatment phase for 3 of the 4 subjects. Only 3 patients provided follow up samples. There is missing data for 1 patient at week 10 and 22.
Measure: Mean (Standard Deviation); unit: RU/mL
Arm/Group | TIO Subjects Who Received BGJ398 (Single Arm)
Number analyzed (Participants) | 4
RU/mL
  Baseline | 814 (911)
  2 Weeks | 213 (158)
  4 Weeks | 330 (87)
  6 Weeks | 229 (123)
  8 Weeks | 304 (154)
  10 Weeks: number analyzed (Participants) | 3
  10 Weeks | 2225 (2015)
  12 Weeks | 430 (409)
  14 Weeks | 270 (65)
  16 Weeks | 360 (75)
  18 Weeks | 185 (151)
  20 Weeks | 274 (118)
  22 Weeks: number analyzed (Participants) | 3
  22 Weeks | 368 (272)
  24 Weeks | 463 (102)
  Follow up | 1568 (1863)

15. Secondary Outcome: Blood Phosphate Levels
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | TIO Subjects Who Received BGJ398 (Single Arm)
Number analyzed (Participants) | 4
mg/dL
  Baseline | 1.6 (0.3)
  Week 2 | 2.7 (0.9)
  Week 4 | 2.9 (1)
  Week 6 | 3.2 (1.3)
  Week 8 | 3.6 (1.5)
  Week 10: number analyzed (Participants) | 3
  Week 10 | 3.1 (0.7)
  Week 12 | 2.9 (1.2)
  Week 14 | 2.8 (1.2)
  Week 16 | 3.4 (1.6)
  Week 18 | 2.5 (0.2)
  Week 20 | 3.0 (1.3)
  Week 22: number analyzed (Participants) | 3
  Week 22 | 3.3 (2.8)
  Week 24 | 3.0 (1.2)
  Follow up | 2.3 (0.4)

16. Secondary Outcome: Blood 1,25-(OH)2-Vitamin D Level
Time Frame: as for outcome 5
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | TIO Subjects Who Received BGJ398 (Single Arm)
Number analyzed (Participants) | 4
pg/mL
  Baseline | 22.5 (16.1)
  Week 2 | 112.3 (94.5)
  Week 4 | 79 (68.4)
  Week 6 | 202.8 (246.5)
  Week 8 | 64.7 (30.7)
  Week 10: number analyzed (Participants) | 3
  Week 10 | 85.7 (63.8)
  Week 12 | 96.5 (61.4)
  Week 14 | 59.8 (28.9)
  Week 16 | 36 (6.1)
  Week 18 | 86.5 (56.3)
  Week 20 | 33 (12.1)
  Week 22: number analyzed (Participants) | 3
  Week 22 | 22.5 (19.1)
  Week 24 | 80.3 (35.7)
  Follow up: number analyzed (Participants) | 3
  Follow up | 51 (32.2)

17. Secondary Outcome: Blood Alkaline Phosphatase
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | TIO Subjects Who Received BGJ398 (Single Arm)
Number analyzed (Participants) | 4
IU/L
  Baseline | 132 (52.3)
  Week 2 | 178.8 (50.7)
  Week 4 | 186.5 (42.1)
  Week 6 | 198 (36.6)
  Week 8 | 171.8 (26.6)
  Week 10: number analyzed (Participants) | 3
  Week 10 | 181.3 (22)
  Week 12 | 170 (18.4)
  Week 14 | 188.3 (29.4)
  Week 16 | 175.5 (14.3)
  Week 18 | 183 (40.4)
  Week 20 | 190.3 (33.6)
  Week 22: number analyzed (Participants) | 3
  Week 22 | 200.7 (48)
  Week 24 | 192.3 (67.4)
  Follow up | 185.7 (17)

18. Secondary Outcome: Tubular Reabsorption of Phosphate
Description: Tubular Reabsorption of Phosphate was calculated using blood phosphate and creatinine, as well as either 24 hour urine or spot urine samples.
Time Frame: as for outcome 13
Population: There were dose interruptions throughout the 24 week treatment phase for 3 of the 4 subjects. Missing urine samples resulted in several time points having fewer than 4 subjects.
Measure: Mean (Standard Deviation); unit: % Filtered Phosphate
Arm/Group | TIO Subjects Who Received BGJ398 (Single Arm)
Number analyzed (Participants) | 4
% Filtered Phosphate
  Baseline | 67 (20)
  Week 2: number analyzed (Participants) | 3
  Week 2 | 82 (13)
  Week 4: number analyzed (Participants) | 3
  Week 4 | 79 (14)
  Week 6 | 84 (14)
  Week 8 | 78 (19)
  Week 10: number analyzed (Participants) | 2
  Week 10 | 50 (36)
  Week 12: number analyzed (Participants) | 3
  Week 12 | 45 (36)
  Week 14 | 82 (15)
  Week 16 | 81 (15)
  Week 18: number analyzed (Participants) | 3
  Week 18 | 77 (13)
  Week 20 | 75 (12)
  Week 22: number analyzed (Participants) | 2
  Week 22 | 81 (11)
  Week 24 | 74 (19)

19. Secondary Outcome: Tubular Maximum Reabsorption Rate of Phosphate to Glomerular Filtration Rate (TmP/GFR)
Description: Tubular maximum reabsorption rate of phosphate to glomerular filtration rate (TmP/GFR) was calculated using blood phosphate and creatinine, as well as either 24 hour urine or spot urine samples.
Time Frame: as for outcome 13
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | TIO Subjects Who Received BGJ398 (Single Arm)
Number analyzed (Participants) | 4
mg/dL
  Baseline | 1.1 (0.5)
  Week 2: number analyzed (Participants) | 3
  Week 2 | 2.5 (1.2)
  Week 4: number analyzed (Participants) | 3
  Week 4 | 2.3 (1.3)
  Week 6 | 3.5 (2.2)
  Week 8 | 3.4 (2.3)
  Week 10: number analyzed (Participants) | 2
  Week 10 | 1.32 (0.9)
  Week 12: number analyzed (Participants) | 3
  Week 12 | 1.52 (1.86)
  Week 14 | 2.76 (1.61)
  Week 16 | 3.44 (2.47)
  Week 18 | 1.98 (0.34)
  Week 20 | 2.31 (1.25)
  Week 22 | 3.86 (2.99)
  Week 24 | 2.61 (1.87)

20. Secondary Outcome: Radiographic Evidence of Tumor-Induced Osteomalacia
Description: In patients with radiographic evidence of TIO, 18FDG PET scans were performed
Time Frame: Baseline and at 24 weeks
Measure: Mean (Standard Deviation); unit: Units
Groups:
- TIO Subjects With Radiographic Evidence of TIO Who Received BGJ398 (Single Arm): TIO subjects with radiographic evidence of TIO were treated with BGJ398 for 24 weeks with optional extension phase. FDG-PET imaging was performed at baseline and at week 24.
Arm/Group | TIO Subjects With Radiographic Evidence of TIO Who Received BGJ398 (Single Arm)
Number analyzed (Participants) | 2
Units
  Baseline SUVmax Tumor | 7.9 (1.3)
  24 Week SUVmax tumor | 3.9 (1.3)

ADVERSE EVENTS:
Time Frame: Patients were monitored for adverse events during 24 weeks of treatment followed by 3 month follow-up period, with optional extension phase up to 37 weeks. If a patient was withdrawn from the study, adverse event data was no longer collected. Subjects who required permanent discontinuation of BGJ398 therapy due to an adverse event continued to be followed in the study until the toxicity had resolved or up to 30 days after study drug discontinuation.
Description: Adverse Events information was collected through investigator assessment every 4 weeks and labs every 2 weeks while on treatment. During the extension phase, adverse event information was collected through investigator and lab assessment every 4 weeks.
Arm/Group | TIO Subjects Who Received BGJ398 (Single Arm)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TIO Subjects Who Received BGJ398 (Single Arm) (N=4)
Anemia (Blood and lymphatic system disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 1
Hearing impairment (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 4
Dry eye (Eye disorders) | 3
Corneal inflamation/keratitis (Eye disorders) | 4
Nuclear Sclerosis (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Hypertrichosis of eyelashes (Ear and labyrinth disorders) | 2
Rash, pustular (Infections and infestations) | 2
C. difficile colitis (Infections and infestations) | 1
Pelvic Infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 3
Neutrophil count decreased (Investigations) | 1
Parathyroid hormone increased (Investigations) | 3
Creatinine increased (Investigations) | 1
Hypercalcemia (Investigations) | 1
Hypercalciuria (Investigations) | 1
Hyperphosphatemia (Investigations) | 3
Weight loss (Investigations) | 1
Vomiting (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Mucositis (Gastrointestinal disorders) | 2
Dysgeusia (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Gastroesophageal reflux (Gastrointestinal disorders) | 1
Pain, musculoskeletal (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry lips (Skin and subcutaneous tissue disorders) | 1
Pain, nails (Skin and subcutaneous tissue disorders) | 4
Nail change/separation (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
This study was terminated early due to a lack of efficacy in the first 4 patients and an unexpectedly high rate of ocular adverse events. As a result, only 4 patients were enrolled in this study. Because of the small sample size, we were unable to perform the planned statistical analysis, and instead the results are primarily descriptive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT03510455/Prot_SAP_000.pdf